CLINICAL TRIAL: NCT06241118
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, 3-arm, Multinational, Multicenter Study to Evaluate the Efficacy and Safety of Amlitelimab by Subcutaneous Injection in Participants Aged 12 Years and Older With Moderate-to-severe Atopic Dermatitis (AD) Who Are on Background Topical Corticosteroids and Have Had an Inadequate Response to Prior Biologic Therapy or Oral Janus Kinase (JAK) Inhibitor Treatment
Brief Title: A Study to Evaluate the Efficacy and Safety of Subcutaneous Amlitelimab on Background Topical Corticosteroids Therapy in Participants Aged 12 Years and Older With Moderate-to-severe AD Who Have Had an Inadequate Response to Prior Biologic Therapy or an Oral JAK Inhibitor
Acronym: AQUA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17599; 2023-508099-12 (Registry Identifier: CTIS); U1111-1295-3059 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Adrenal Cortex Hormones; Tacrolimus; pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Amlitelimab dose 1 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab; Drug: Topical corticosteroids; Drug: Topical tacrolimus or pimecrolimus
- Amlitelimab dose 2 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab; Drug: Topical corticosteroids; Drug: Topical tacrolimus or pimecrolimus
- Placebo (Placebo Comparator): Subcutaneous injection as per protocol
  Interventions: Drug: Placebo; Drug: Topical corticosteroids; Drug: Topical tacrolimus or pimecrolimus

INTERVENTIONS:
Drug: Amlitelimab — Pharmaceutical form: Injection solution Route of administration: Subcutaneous
  Other Names: SAR445229
  Arms: Amlitelimab dose 1; Amlitelimab dose 2
Drug: Placebo — Pharmaceutical form: Injection solution Route of administration: Subcutaneous
  Arms: Placebo
Drug: Topical corticosteroids — Pharmaceutical form: Various Topical formulation Route of administration: Topical
Drug: Topical tacrolimus or pimecrolimus — Pharmaceutical form: Various Topical formulation Route of administration: Topical

SUMMARY:
This is a parallel group, Phase 3, multinational, multicenter, randomized, double-blind, placebo-controlled, 3-arm study for treatment of participants diagnosed with moderate-to-severe AD on background TCS who have had inadequate response to prior biologic or oral JAKi therapy.

The purpose of this study is to measure the efficacy and safety of treatment with amlitelimab solution for subcutaneous (SC) injection compared with placebo in participants with moderate-to-severe AD aged 12 years and older on background TCS and have had an inadequate response to prior biologic or an oral JAKi therapy.

Study details include:

At the end of the treatment period, participants will have the option to enter the Long-Term Safety Study LTS17367 (RIVER-AD).

The study duration will be up to 56 weeks for participants not entering the long-term safety study (LTS17367 [RIVER-AD]) including a 2 to 4-week screening, a 36-week randomized double-blind period, and a 16-week safety follow-up.

The study duration will be up to 40 weeks for participants entering the long-term safety study (LTS17367 [RIVER-AD]) including a 2 to 4-week screening and a 36-week randomized double-blind period.

The total treatment duration will be up to 36 weeks. The total number of visits will be up to 13 visits (or 12 visits for those entering the long-term safety study LTS17367 [RIVER-AD] study).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 12 years of age (when signing informed consent form)
* Diagnosis of AD for at least 1 year (defined by the American Academy of Dermatology Consensus Criteria)
* Documented history prior to screening visit of inadequate response to a biologic AD medication or an oral JAKi therapy.
* v-IGA-AD of 3 or 4 at baseline visit
* EASI score of 16 or higher at baseline
* AD involvement of 10% or more of BSA at baseline
* Weekly average of daily PP-NRS of ≥ 4 at baseline visit.
* Able and willing to comply with requested study visits and procedures
* Body weight ≥25 kg

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Skin co-morbidity that would adversely affect the ability to undertake AD assessments
* Known history of or suspected significant current immunosuppression
* Any malignancies or history of malignancies prior to baseline (with the exception of non-melanoma skin cancer excised and cured >5 years prior to baseline)
* History of solid organ or stem cell transplant
* Any active or chronic infection including helminthic infection requiring systemic treatment within 4 weeks prior to baseline
* Positive for human immunodeficiency virus (HIV), Hepatitis B or hepatitis C at screening visit
* Having active tuberculosis (TB), latent TB, a history of incompletely treated TB, suspected extrapulmonary TB infection, or who are at high risk of contracting TB
* Having received any of the specified therapy within the specified timeframe(s) prior to the baseline visit
* In the Investigator's opinion, any clinically significant laboratory results or protocol specified laboratory abnormalities at screening
* History of hypersensitivity or allergy to any of the excipients or investigational medicinal product (IMP)

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-09-14 (Estimated)

PRIMARY OUTCOMES:
EU, EU reference countries, and Japan: Proportion of participants with Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) of 0 (clear) or 1 (almost clear) and a reduction from baseline of ≥2 points at Week 36 | Week 36
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
EU, EU reference countries, and Japan: Proportion of participants reaching 75% reduction from baseline in Eczema Area and Severity Index (EASI) score (EASI75) at Week 36 | Week 36
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
US and US reference countries: Proportion of participants with vIGA-AD of 0 (clear) or 1 (almost clear) and a reduction from baseline of ≥2 points at Week 36 | Week 36
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).

SECONDARY OUTCOMES:
Proportion of participants reaching EASI-75 at Week 36 (for US and US reference countries only) | Week 36
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score.
Proportion of participants with vIGA-AD 0 (clear) or 1 (almost clear) with presence of only barely perceptible erythema (no induration/papulation, no lichenification, no oozing or crusting and a reduction from baseline of ≥2 points) | Baseline to Week 36
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants with ≥4-point reduction in weekly average of daily Peak Pruritus-Numerical Rating Scale (PP-NRS) from baseline in participants with baseline weekly average of daily PP-NRS ≥4 | Baseline to Week 36
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Proportion of participants reaching EASI-75 | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score.
Proportion of participants with vIGA-AD of 0 (clear) or 1 (almost clear) and a reduction from baseline of ≥2 points | Baseline to Week 24
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants reaching EASI-90 | Baseline to Week 36
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-90 is 90% reduction from baseline in EASI score.
Proportion of participants reaching EASI-100 | Baseline to Week 36
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-100 is 100% reduction from baseline in EASI score.
Proportion of participants with PP-NRS ≤1 | Baseline to Week 36
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Change in Dermatology Life Quality Index (DLQI) from baseline in participants with age ≥16 years old | Baseline to Week 36
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Proportion of participants with a reduction in DLQI ≥4 from baseline in participants with age ≥16 years old and with DLQI baseline ≥4 | Baseline to Week 36
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Change in Children Dermatology Life Quality Index (CDLQI) from baseline in participants with age ≥12 to <16 years | Baseline to Week 36
  The CDLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in children aged 4-<16 years. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Proportion of participants with a reduction in CDLQI ≥6 from baseline in participants with age ≥12 to <16 years old and with CDLQI baseline ≥6 | Baseline to Week 36
  The CDLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in children aged 4-<16 years. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Change in Hospital Anxiety Depression Scale (HADS) from baseline | Baseline to Week 36
  The HADS is 14-item questionnaire with two subscales: anxiety & depression. Each subscale (anxiety & depression) ranges 0-21. The total HADS score ranges 0-42 with higher score indicating a poorer state.
Proportion of participants with HADS subscale Anxiety (HADS-A) <8 in participants with baseline HADS-A ≥8 | Baseline to Week 36
  HADS-A score ranges 0-21 with higher score indicating a poorer state.
Proportion of participants with HADS subscale Depression (HADS-D) <8 in participants with HADS-D baseline ≥8 | Baseline to Week 36
  HADS-D score ranges 0-21 with higher score indicating a poorer state.
Absolute change in weekly average of daily Skin Pain-Numerical Rating Scale (SP-NRS) from baseline | Baseline to Week 36
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Proportion of participants with a reduction in weekly average of daily SP-NRS ≥4 from baseline in participants with baseline weekly average of daily SP-NRS ≥4 | Baseline to Week 36
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Percent change in weekly average of daily SP-NRS from baseline | Baseline to Week 36
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Proportion of participants with vIGA-AD 0 (clear) | Baseline to Week 36
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Absolute change in weekly average of daily Sleep Disturbance-Numerical Rating Scale (SD-NRS) from baseline | Baseline to Week 36
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Proportion of participants with a reduction in weekly average of daily SD-NRS ≥3 from baseline in participants with Baseline weekly average of daily SD-NRS ≥3 | Baseline to Week 36
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Percent change in weekly average of daily SD-NRS | Baseline to Week 36
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Percent change in EASI score from baseline | Baseline to Week 36
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Percent change in weekly average of daily PP-NRS from baseline | Baseline to Week 36
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Absolute change in weekly average of daily PP-NRS from baseline | Baseline to Week 36
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Proportion of participants reaching EASI-50 | Baseline to Week 36
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-50 is 50% reduction from baseline in EASI score.
Proportion of participants with EASI ≤7 | Baseline to Week 36
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Change in percent Body Surface Area (BSA) affected by AD from baseline | Baseline to Week 36
Percent change in Scoring Atopic Dermatitis (SCORAD) index from baseline | Baseline to Week 36
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Absolute change in SCORAD index from baseline | Baseline to Week 36
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Proportion of participants with a reduction in SCORAD ≥ 8.7 points from baseline in participants with baseline SCORAD score ≥ 8.7 | Baseline to Week 36
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Proportion of participants with a reduction in Patient Oriented Eczema Measure (POEM) ≥4 from baseline in participants with POEM Baseline ≥4 | Baseline to Week 36
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a 5-point scale; 0 (no days) to 4 (every day in the last week). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (very severe). Higher scores indicated more severe disease and poor quality of life.
Change in POEM from baseline | Baseline to Week 36
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a 5-point scale; 0 (no days) to 4 (every day in the last week). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (very severe). Higher scores indicated more severe disease and poor quality of life.
Proportion of participants with rescue medication use | Baseline to Week 36
Time to onset of effect on PP-NRS as measured by proportion of participants with an improvement (reduction) in PP-NRS by ≥4 | Baseline to Week 36
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Percentage of TCS/TCI free days | Baseline to Week 36
Percentage of participants who experienced Treatment-Emergent Adverse Events (TEAEs), experienced Treatment-Emergent Serious Adverse Events (TESAEs) and/or Treatment-Emergent Adverse Events of Special Interest (AESI) | Baseline to Week 52
Serum amlitelimab concentrations | Baseline to Week 52
Incidence of antidrug antibodies (ADAs) of amlitelimab | Baseline to Week 52
Time to onset of effect on vIGA-AD as measured by proportion of participants with vIGA-AD 0 (clear) or 1 (almost clear) and a reduction from baseline ≥2 during the 36-week treatment period | Baseline to Week 36
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Time to onset of effect on EASI as measured by proportion of participants reaching a 75% reduction from baseline in EASI score during the 36-week treatment period | Baseline to Week 36
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score.

CONTACTS AND LOCATIONS:
Locations (148):
- United States (42):
  - University of Alabama at Birmingham- Site Number : 8401267, Birmingham, Alabama
  - Center for Dermatology and Plastic Surgery- Site Number : 8401119, Scottsdale, Arizona
  - Arkansas Dermatology- Site Number : 8401244, Little Rock, Arkansas
  - Encino Research Center- Site Number : 8401042, Encino, California
  - Center for Dermatology Clinical Research- Site Number : 8401018, Fremont, California
  - Long Beach Clinical Trials- Site Number : 8401188, Long Beach, California
  - Dermatology Research Associates - Los Angeles- Site Number : 8401092, Los Angeles, California
  - LA Universal Research Center- Site Number : 8401064, Los Angeles, California
  - University Dermatology Trials- Site Number : 8401339, Newport Beach, California
  - Rady Children's Hospital- Site Number : 8401291, San Diego, California
  - Therapeutics Clinical Research- Site Number : 8401283, San Diego, California
  - Paradigm Clinical Research - Wheat Ridge- Site Number : 8401245, Wheat Ridge, Colorado
  - Encore Medical Research of Boynton Beach- Site Number : 8401030, Boynton Beach, Florida
  - St. Jude Clinical Research- Site Number : 8401287, Doral, Florida
  - Apex Clinical Research - Jacksonville- Site Number : 8401332, Jacksonville, Florida
  - Global Clinical Professionals (GCP)- Site Number : 8401045, St. Petersburg, Florida
  - Avita Clinical Research- Site Number : 8401073, Tampa, Florida
  - Northwestern University- Site Number : 8401285, Chicago, Illinois
  - NorthShore University Health System - Endeavor Health Medical Group - Skokie - Woods Drive- Site Number : 8401038, Skokie, Illinois
  - Dawes Fretzin Clinical Research- Site Number : 8401015, Indianapolis, Indiana
  - Equity Medical - Bowling Green- Site Number : 8401296, Bowling Green, Kentucky
  - Tandem Clinical Research - Metairie- Site Number : 8401187, Metairie, Louisiana
  - University of Michigan Health System - Ann Arbor- Site Number : 8401290, Ann Arbor, Michigan
  - MI Skin Center- Site Number : 8401307, Northville, Michigan
  - Skin Specialists- Site Number : 8401068, Omaha, Nebraska
  - Schweiger Dermatology Group - East Windsor- Site Number : 8401338, East Windsor, New Jersey
  - The University of New Mexico- Site Number : 8401263, Albuquerque, New Mexico
  - Equity Medical- Site Number : 8401239, New York, New York
  - Sadick Research Group - New York - Park Avenue- Site Number : 8401050, New York, New York
  - Cincinnati Children's Hospital Medical Center- Site Number : 8401279, Cincinnati, Ohio
  - Oregon Health & Science University (OHSU)- Site Number : 8401247, Portland, Oregon
  - Paddington Testing Company- Site Number : 8401041, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia- Site Number : 8401193, Philadelphia, Pennsylvania
  - Medical University of South Carolina - Charleston - Jonathan Lucas Street- Site Number : 8401282, Charleston, South Carolina
  - Arlington Research Center- Site Number : 8401248, Arlington, Texas
  - McGovern Medical School - UT Physicians Dermatology - Bellaire Station- Site Number : 8401288, Bellaire, Texas
  - Reveal Research Institute - Dallas- Site Number : 8401219, Dallas, Texas
  - Advanced Research Institute - Odgen- Site Number : 8401057, Ogden, Utah
  - Virginia Dermatology & Skin Cancer Center- Site Number : 8401047, Norfolk, Virginia
  - North Sound Dermatology- Site Number : 8401280, Mill Creek, Washington
  - Children's Wisconsin- Site Number : 8401246, Milwaukee, Wisconsin
  - Cheyenne Skin Clinic- Site Number : 8401234, Cheyenne, Wyoming
- Argentina (4):
  - Investigational Site Number : 0320007, Rosario, Santa Fe Province
  - Investigational Site Number : 0320011, Buenos Aires
  - Investigational Site Number : 0320019, Buenos Aires
  - Investigational Site Number : 0320014, Córdoba
- Australia (2):
  - Investigational Site Number : 0360008, Melbourne, Victoria
  - Investigational Site Number : 0360006, Melbourne, Victoria
- Brazil (6):
  - Centro de Pesquisas da Clínica IBIS- Site Number : 0760002, Salvador, Estado de Bahia
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre- Site Number : 0760005, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC- Site Number : 0760001, Santo André, São Paulo
  - Clinica de Alergia Martti Antila- Site Number : 0760006, Sorocaba, São Paulo
  - Hospital Alemao Oswaldo Cruz - São Paulo- Site Number : 0760010, São Paulo
  - Centro de Desenvolvimento em Estudos ClÌnicos Brasil- Site Number : 0760014, São Paulo
- Canada (7):
  - Investigational Site Number : 1240019, Calgary, Alberta
  - Investigational Site Number : 1240016, Edmonton, Alberta
  - Investigational Site Number : 1240058, Burlington, Ontario
  - Investigational Site Number : 1240020, Hamilton, Ontario
  - Investigational Site Number : 1240053, London, Ontario
  - Investigational Site Number : 1240054, Toronto, Ontario
  - Investigational Site Number : 1240028, Regina, Saskatchewan
- Chile (5):
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520010, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
- China (13):
  - Investigational Site Number : 1560031, Changchun
  - Investigational Site Number : 1560021, Guangzhou
  - Investigational Site Number : 1560036, Guangzhou
  - Investigational Site Number : 1560044, Hangzhou
  - Investigational Site Number : 1560002, Hangzhou
  - Investigational Site Number : 1560009, Hangzhou
  - Investigational Site Number : 1560034, Nanyang
  - Investigational Site Number : 1560024, Ningbo
  - Investigational Site Number : 1560035, Ningbo
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560041, Shenyang
  - Investigational Site Number : 1560038, Wuhan
  - Investigational Site Number : 1560032, Xi'an
- France (6):
  - Investigational Site Number : 2500011, Bordeaux
  - Investigational Site Number : 2500014, Clermont-Ferrand
  - Investigational Site Number : 2500004, Créteil
  - Investigational Site Number : 2500001, Lille
  - Investigational Site Number : 2500017, Paris
  - Investigational Site Number : 2500012, Rouen
- Germany (6):
  - Investigational Site Number : 2762203, Berlin
  - Investigational Site Number : 2762202, Blankenfelde-Mahlow
  - Investigational Site Number : 2761001, Dresden
  - Investigational Site Number : 2760022, Frankfurt
  - Investigational Site Number : 2761002, Lübeck
  - Investigational Site Number : 2760019, Witten
- Greece (4):
  - Investigational Site Number : 3000004, Athens
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000005, Athens
  - Investigational Site Number : 3000002, Thessaloniki
- Israel (3):
  - Investigational Site Number : 3760005, Beersheba
  - Investigational Site Number : 3760008, Ramat Gan
  - Investigational Site Number : 3760007, Tel Aviv
- Italy (5):
  - Investigational Site Number : 3800017, Naples, Napoli
  - Investigational Site Number : 3800020, Turin, Torino
  - Investigational Site Number : 3800016, Chieti
  - Investigational Site Number : 3800021, Modena
  - Investigational Site Number : 3800015, Perugia
- Japan (6):
  - Investigational Site Number : 3923113, Yokohama, Kanagawa
  - Investigational Site Number : 3923109, Habikino, Osaka
  - Investigational Site Number : 3923110, Sakai, Osaka
  - Investigational Site Number : 3923106, Mibu, Tochigi
  - Investigational Site Number : 3920001, Tachikawa, Tokyo
  - Investigational Site Number : 3920007, Hiroshima
- Mexico (2):
  - Investigational Site Number : 4840011, Monterrey, Nuevo León
  - Investigational Site Number : 4840003, Veracruz
- Investigational Site Number : 5280001, Utrecht, Netherlands
- Poland (5):
  - Investigational Site Number : 6162417, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160002, Lublin, Lublin Voivodeship
  - Investigational Site Number : 6162411, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160001, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160006, Gdansk, Pomeranian Voivodeship
- Investigational Site Number : 2500016, Saint-Pierre, Reunion
- Investigational Site Number : 6820001, Riyadh, Saudi Arabia
- South Korea (5):
  - Investigational Site Number : 4100002, Ansan-si, Gyeonggi-do
  - Investigational Site Number : 4100014, Seongnam-si, Gyeonggi-do
  - Investigational Site Number : 4100015, Bupyeong-gu, Incheon-gwangyeoksi
  - Investigational Site Number : 4100007, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
- Spain (6):
  - Investigational Site Number : 7240002, Badalona, Barcelona [Barcelona]
  - Investigational Site Number : 7240017, Majadahonda, Madrid
  - Investigational Site Number : 7240016, Pozuelo de Alarcón, Madrid
  - Investigational Site Number : 7240020, Seville, Sevilla
  - Investigational Site Number : 7242505, Alicante
  - Investigational Site Number : 7242503, Madrid
- Taiwan (4):
  - Investigational Site Number : 1583201, Kaohsiung City
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1580003, Taipei
  - Investigational Site Number : 1583203, Taoyuan
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920008, Gaziantep
  - Investigational Site Number : 7920005, Istanbul
  - Investigational Site Number : 7920002, Istanbul
- United Arab Emirates (3):
  - Investigational Site Number : 7841002, Abu Dhabi
  - Investigational Site Number : 7840001, Abu Dhabi
  - Investigational Site Number : 7840002, Abu Dhabi
- United Kingdom (8):
  - Investigational Site Number : 8260013, Bristol, Bristol, City of
  - Investigational Site Number : 8260012, Plymouth, Devon
  - Investigational Site Number : 8262603, London, England
  - Investigational Site Number : 8260015, London, England
  - Investigational Site Number : 8260003, Portsmouth, Hampshire
  - Investigational Site Number : 8260009, Leeds, North Yorkshire
  - Investigational Site Number : 8260010, Nottingham, Nottinghamshire
  - Investigational Site Number : 8260008, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17599 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25595&tenant=MT_SNY_9011